CLINICAL TRIAL: NCT07394998
Title: Comparison of Exercise Capacity, Muscle Oxygenation and Aortic Stiffness in Patients With a History of Mitral Valve Intervention for Mitral Stenosis With Healthy Subjects
Brief Title: Assessment of Exercise Capacity, Muscle Oxygenation and Aortic Stiffness in Patients With Mitral Stenosis
Status: Recruiting | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: 2024 1390
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Mitral Stenosis
Keywords: cardiopulmonary exercise test; aortic stiffness; muscle oxygenation; physical activity; mitral stenosis
MeSH Terms: conditions — Mitral Valve Stenosis; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients group: This group includes patients who have undergone mitral stenosis intervention for mitral stenosis. Patients exercise capacity using Cardiopulmonary Exercise Test (CPET), muscle oxygenation with a near-infrared spectroscopy device, respiratory functions with a spirometer, respiratory muscle strength with a mouth pressure measurement device, respiratory muscle endurance with an incremental threshold loading respiratory muscle endurance test, aortic stiffness with an arteriograph, physical activity level with a multisensor physical activity monitor and quality of life with the SF-36 Short Form will be evaluated.
- Healthy Controls Group: Healthy controls will be evaluated for exercise capacity with the Cardiopulmonary Exercise Test (CPET), muscle oxygenation with a near-infrared spectroscopy device, respiratory functions with a spirometer, respiratory muscle strength with a mouth pressure measurement device, respiratory muscle endurance with an incremental threshold loading respiratory muscle endurance test, aortic stiffness with an arteriograph, physical activity level with a multisensor physical activity monitor, and quality of life with the SF-36 Short Form.

SUMMARY:
Heart valve diseases are the most common cause of mortality and morbidity after coronary artery disease, hypertension, and heart failure. In patients with mitral stenosis, the narrowed valve restricts blood flow, causing symptoms such as shortness of breath, fatigue, exertional dyspnea, orthopnea, and paroxysmal nocturnal dyspnea. These patients may experience decreased exercise capacity and physical activity levels, deterioration in quality of life, and deterioration in respiratory function. When reviewing the literature, we see that the study groups evaluating these factors are generally not homogeneous, and most studies conducted in patients with mitral stenosis evaluate patients who have undergone percutaneous mitral balloon valvuloplasty.

DETAILED DESCRIPTION:
In mitral valve stenosis, blood flow from the left atrium to the left ventricle is mechanically restricted, resulting in increased pressure in the left atrium, pulmonary vascular bed, and right chambers of the heart. The narrowed mitral valve obstructs the flow of blood from the lungs to the heart, causing shortness of breath in patients. Increased blood volume in the left atrium may cause palpitations. Other symptoms include fatigue, exertional dyspnea, orthopnea, paroxysmal nocturnal dyspnea, chest pain, and dizziness.

Patients with mitral stenosis are expected to have decreased exercise capacity due to restrictive lung function, chronotropic insufficiency, limited stroke volume, and the effects of peripheral factors. Studies evaluating the exercise capacity of patients who have undergone surgery for mitral stenosis are limited.

After cardiac surgery, oxygen saturation decreases in the acute period, and hemodynamic and systemic oxygenation are often impaired. It has been suggested that muscle deoxygenation may also occur in patients with mitral stenosis due to these reasons. Studies investigating skeletal muscle oxygenation after mitral valve surgery are limited in the literature. While surgery for heart valve lesions improves cardiac function, changes in the thoracic compartment are major causes of mortality and morbidity. These changes reduce cardiorespiratory capacity, leading to physical inactivity, loss of muscle strength, and loss of fitness in patients.

Inspiratory muscle performance is impaired in patients who have undergone valve replacement surgery. Better inspiratory muscle performance in these patients is associated with better physical function. This relationship between respiratory muscle strength and exercise capacity demonstrates the importance of assessing respiratory muscle strength. Mitral valve stenosis is associated with impaired aortic stiffness. In patients with heart failure, aortic stiffening plays a role in hemodynamic deterioration due to its adverse effect on left ventricular function and coronary artery perfusion. In conclusion, aortic stiffness has been shown to exacerbate the disease through multiple mechanisms. Inadequate physical activity after heart valve surgery is associated with a higher mortality rate, while adequate physical activity prevents cardiovascular events and reduces mortality in the long term. Physical activity is an important prognostic factor in patients who have undergone cardiac surgery. The quality of life of patients improves after heart valve surgery. The extent of improvement may vary depending on the surgical method used.

The primary objective of the study is to compare exercise capacity, muscle oxygenation, aortic stiffness, and quality of life in patients who have undergone surgery for mitral stenosis with those in healthy individuals.

The secondary objective of the study is to compare respiratory muscle strength and endurance, pulmonary function, and physical activity levels in patients who have undergone surgery for mitral stenosis with those in healthy individuals.

Primary outcomes are exercise capacity, muscle oxygenation, aortic stiffness, and quality of life.

Secondary outcomes are respiratory muscle strength, respiratory muscle endurance, pulmonary function and physical activity level.

ELIGIBILITY:
Inclusion Criteria:

Patients;

* Between the ages of 18-80
* Patients who have undergone mitral valve intervention due to mitral stenosis
* At least 3 months have passed since the intervention

Healthy controls;

* Between the ages of 18 and 80
* Agreeing to participate voluntarily in the study

Exclusion Criteria:

Patients;

* Patients who have undergone aortic valve intervention other than mitral valve intervention
* Acute infection
* Orthopedic, neurological or psychological disorders that will affect functional capacity

Healthy Controls;

* diagnosed chronic disease,
* acute infection
* A smoking history of at least 10 packs×years or more

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients with a history of mitral valve intervention for mitral stenosis and 30 healthy individuals will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Maximal Exercise Capacity | Through study completion, an average of 1 year
  Maximal Exercise capacity will be evaluated with Cardiopulmonary Exercise testing. The Cardiopulmonary Exercise Testing will be applied according to American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Muscle Oxygenation | Through study completion, an average of 1 year
  Peripheral muscle oxygen will be measured by near-infrared spectrometry. The device probes will be placed on the trunk and lower extremities. The device allows to display of the percentage of oxygen, the concentration of oxyhemoglobin, and deoxyhemoglobin, the difference between oxyhemoglobin and deoxyhemoglobin, and the total hemoglobin. These parameters will be evaluated in our study.
Aortic Stiffness | Through study completion, an average of 1 year
  Aortic stiffness will be assessed non-invasively using the SphygmoCor XCEL® device, whose validity and reliability have been proven. The device measures carotid-femoral pulse wave velocity (cfPWV).
Quality of Life (Short Form 36) | through study completion, an average of 1 year
  Health-related quality of life will be assessed using the valid and reliable Short Form 36 (SF-36). The SF-36 consists of a total of 36 items across 8 health domains. The 8 health domains assessed are general health, physical functioning, social functioning, physical limitations due to health problems, emotional limitations due to health problems, pain, mental health, and energy/vitality. It assesses the individual's last month using a Likert scale. Each health domain is scored between 0 and 100. A higher score indicates better health status.

SECONDARY OUTCOMES:
Respiratory Muscle Strength | Through study completion, an average of 1 year
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength were measured using a portable mouth pressure measuring device according to American Thoracic Society and European Respiratory Society criteria.
Respiratory Muscle Endurance | Through study completion, an average of 1 year
  Respiratory muscle endurance will be assessed using the incremental threshold loading test.
Pulmonary Function (Forced vital capacity (FVC)) | Through study completion, an average of 1 year
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, forced vital capacity (FVC)was evaluated.
Pulmonary Function (Forced expiratory volume in first second (FEV1)) | Through study completion, an average of 1 year
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, forced expiratory volume in first second (FEV1) was evaluated.
Pulmonary Function (FEV1/FVC) | Through study completion, an average of 1 year
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, FEV1/FVC was evaluated.
Pulmonary Function (Flow rate 25-75% of forced expiratory volume (FEF25-75%)) | Through study completion, an average of 1 year
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, Flow rate 25-75% of forced expiratory volume (FEF25-75%)was evaluated.
Pulmonary Function (Peak flow rate (PEF)) | Through study completion, an average of 1 year
  Pulmonary function was evaluated using the spirometry. Dynamic lung volume measurements were conducted according to ATS and ERS criteria. With the device, peak flow rate (PEF) was evaluated.
Physical Activity Level | Through study completion, an average of 1 year
  Physical activity level will be assessed using a multi-sensor activity monitor. The patient will wear the multi-sensor activity monitor continuously for 4 days using a belt at hip level on the non-dominant side.

CONTACTS AND LOCATIONS:
Overall Officials: Ebrar TÜLÜMENOĞLU, Pt, Study Chair — Gazi University; Özden SEÇKİN GÖBÜT, Dr, Principal Investigator — Gazi University; Serkan ÜNLÜ, Dr, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Physiotherapy and Rehabilitation, Cardiopulmonary Rehabilitation Unit, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopaschuk GD, Jaswal JS. Hypoxia-induced adaptation to mitral regurgitation: a role for K ATP channel up-regulation? J Am Coll Cardiol. 2012 Jan 24;59(4):397-9. doi: 10.1016/j.jacc.2011.09.056. Epub 2011 Nov 30. No abstract available. PMID 22133354
- [Background] Kopp R, Dommann K, Rossaint R, Schalte G, Grottke O, Spillner J, Rex S, Marx G. Tissue oxygen saturation as an early indicator of delayed lactate clearance after cardiac surgery: a prospective observational study. BMC Anesthesiol. 2015 Oct 30;15:158. doi: 10.1186/s12871-015-0140-7. PMID 26518485
- [Background] Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Feb 2;143(5):e35-e71. doi: 10.1161/CIR.0000000000000932. Epub 2020 Dec 17. PMID 33332149
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Reference Values for Arterial Stiffness' Collaboration. Determinants of pulse wave velocity in healthy people and in the presence of cardiovascular risk factors: 'establishing normal and reference values'. Eur Heart J. 2010 Oct;31(19):2338-50. doi: 10.1093/eurheartj/ehq165. Epub 2010 Jun 7. PMID 20530030
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Inci S, Nar G, Erol MK, Demirelli S, Duman H, Serdar S, Erol F. The effects of successful percutaneous mitral balloon valvuloplasty on acute and intermediate term aortic stiffness. Echocardiography. 2015 May;32(5):813-8. doi: 10.1111/echo.12799. Epub 2014 Oct 27. PMID 25345485
- [Background] Demirbag R, Sade LE, Aydin M, Bozkurt A, Acarturk E. The Turkish registry of heart valve disease. Turk Kardiyol Dern Ars. 2013 Jan;41(1):1-10. doi: 10.5543/tkda.2013.71430. PMID 23518931
- [Background] Laufer-Perl M, Gura Y, Shimiaie J, Sherez J, Pressman GS, Aviram G, Maltais S, Megidish R, Halkin A, Ingbir M, Biner S, Keren G, Topilsky Y. Mechanisms of Effort Intolerance in Patients With Rheumatic Mitral Stenosis: Combined Echocardiography and Cardiopulmonary Stress Protocol. JACC Cardiovasc Imaging. 2017 Jun;10(6):622-633. doi: 10.1016/j.jcmg.2016.07.011. Epub 2016 Nov 16. PMID 27865723
- [Background] van Laar C, TImman ST, Noyez L. Decreased physical activity is a predictor for a complicated recovery post cardiac surgery. Health Qual Life Outcomes. 2017 Jan 7;15(1):5. doi: 10.1186/s12955-016-0576-6. PMID 28069013